CLINICAL TRIAL: NCT02434718
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Aducanumab (BIIB037) in Japanese Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Single and Multiple Ascending Dose Study of Aducanumab (BIIB037) in Japanese Participants With Alzheimer's Disease
Acronym: PROPEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 221AD104
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — aducanumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): IV infusion in cohorts assigned to low dose 1; 1 participant per cohort will receive placebo
  Interventions: Drug: Aducanumab; Drug: Placebo
- Cohort 2 (Experimental): IV infusion in cohorts assigned to low dose 2; 1 participant per cohort will receive placebo
  Interventions: Drug: Aducanumab; Drug: Placebo
- Cohort 3 (Experimental): IV infusion in cohorts assigned to high dose; 1 participant per cohort will receive placebo
  Interventions: Drug: Aducanumab; Drug: Placebo
- Cohort 4 (Experimental): IV infusion in cohorts assigned to mid dose; 1 participant per cohort will receive placebo
  Interventions: Drug: Aducanumab; Drug: Placebo

INTERVENTIONS:
Drug: Aducanumab — As described in the treatment arm
Drug: Placebo — IV administration of 0.9% sodium chloride

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single and multiple intravenous (IV) infusions of Aducanumab in Japanese participants with mild to moderate Alzheimer's Disease (AD). The secondary objectives of this study are as follows: To evaluate the serum pharmacokinetics (PK) of Aducanumab after single and multiple intravenous (IV) infusions of Aducanumab; To evaluate the effect of single and multiple IV infusions of Aducanumab on immunogenicity.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be ambulatory
* Must have a clinical diagnosis of mild to moderate AD
* Must be in good health as determined by the Investigator, based on medical history and Screening assessments
* Must have a caregiver who, understands the study and assents to accompany the subject to all study site visits, provide information to the Investigator/study site staff, specifically about cognitive abilities and AEs/SAEs and return for per-protocol follow-up visits and procedures
* Must consent to blood sample collection for deoxyribonucleic acid (DNA; genotyping) and ribonucleic acid (RNA; for potential future analysis).

Key Exclusion Criteria:

* Any medical or neurological condition (other than AD) that in the opinion of the Investigator could be a contributing cause of the subject's dementia
* Transient ischemic attack or stroke or any unexplained loss of consciousness within 1 year prior to Screening
* Poorly controlled diabetes mellitus, as defined by having dosage adjustment of diabetic medication within the 3 months prior to Day 1
* History of unstable angina, myocardial infarction, chronic heart failure
* Chronic, uncontrolled hypertension
* History of seizure within 3 years prior to Screening
* History within the past 6 months or evidence of clinically significant psychiatric illness
* History of severe allergic or anaphylactic reactions, or history of hypersensitivity to any of the inactive ingredients in the drug product

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of adverse events (AE) / serious adverse events(SAE) | Up to week 42
Clinically significant changes in vital signs and 12-lead electrocardiogram (ECG) data; abnormalities in neurological and physical examinations | Up to week 42
Brain magnetic resonance imaging (MRI) findings to assess amyloid-related imaging abnormalities (ARIA), including incidence of ARIA-E (edema) or ARIA-H (hemosiderosis) | Up to week 42

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) from time zero extrapolated to infinity (AUC0-∞) | Up to 8 weeks post dosing
AUC from time zero to time of the last measurable concentration (AUC0-last) | Up to 8 weeks post dosing
Maximum observed concentration (Cmax) | Up to 8 weeks post dosing
Time to Cmax (Tmax) | Up to 8 weeks post dosing
Elimination half-life (t1/2) | Up to 8 weeks post dosing
Volume of distribution at steady state (Vss) | Up to 8 weeks post dosing
Clearance (CL) after a single IV infusion of aducanumab | Up to 8 weeks post dosing
Incidence of anti-aducanumab antibodies in serum | Up to week 42

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (7):
- Japan (7):
  - Research Site, Tōon, Ehime
  - Research Site, Kobe, Hyōgo
  - Research Site, Kamakura, Kanagawa
  - Research Site, Kanzaki, Saga-ken
  - Research Site, Kodaira, Tokoyo
  - Research Site, Shinjuku, Tokoyo
  - Research Site, Kyoto